CLINICAL TRIAL: NCT05327881
Title: Serum Rennin Kinetics Versus Serum Lactate Kinetics as Predictors of Mortality in Septic Shock Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Rabiee Ali, Assistant Lecturer, Anesthesia and ICU department, Faculty of medicine, Assiut University, Assiut University
Other Study IDs: ReninvsLactate in septic shock
Record Dates: First submitted 2022-03-16; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Septic shock patients: Adult patients on vasopressors for greater than 6 hours to maintain a mean arterial pressure greater than or equal to 65 mm Hg. Inclusion criteria: age over 18, urinary catheter in situ, anticipated stay >24 hours, and signed informed consent by patient or next-of-kin.
  Septic shock was defined as persistent hypotension (defined as the need for vasopressors to maintain mean arterial pressure ≥ 65 mm Hg, and a serum lactate level > 18 mg/dL [2 mmol/L] despite adequate volume resuscitation
  Interventions: Diagnostic Test: Plasma renin concentrations will be measured at enrollment and at 24, 48, and 72 hours. Whole blood lactate measurements will be performed according to normal standard of care.

INTERVENTIONS:
Diagnostic Test: Plasma renin concentrations will be measured at enrollment and at 24, 48, and 72 hours. Whole blood lactate measurements will be performed according to normal standard of care. — Measurement of Whole Blood Lactate Concentrations:
  Whole blood lactate concentrations were measured using ABL 800 series analyzers. The IRB (Institutional Review Board) protocol specified that lactate concentrations could be obtained as part of routine care, but lactate concentrations were not measured independently for research purposes.
  Measurement of Plasma Renin Concentrations:
  Discarded whole blood samples (waste blood samples) in EDTA (ethylenediaminetetraacetic acid) (BD Vacutainer, 4 mL) tubes were prospectively collected from each patient at the time of study enrollment and at 24, 48, and 72 hours.
  Plasma active renin levels were measured using the active renin enzyme-linked immunosorbent assay kit (DRG International, Township, NJ)

SUMMARY:
Whole blood lactate concentration is widely used in shock states to assess perfusion. We aimed to determine if the change in plasma renin concentration over time would be superior to the change in lactate concentration for predicting in-hospital mortality in septic shock patients.

DETAILED DESCRIPTION:
Resuscitation in the ICU was traditionally based on blood pressure (1, 2). An assumption that adequate tissue perfusion cannot be made at pressures of 65 mm Hg, and the number itself has been challenged in other investigations (1, 3, 4). Lactate has long been regarded as an adequate indicator of tissue perfusion and prognosis. Most critical care resuscitation are guided by serial lactate levels as a mean to understand the flow and perfusion side of resuscitative aims (2, 5). Not all high lactate levels are indicators of poor tissue perfusion (6).In 2017, Khanna et al (7) reinvigorated the interest in the renin-angiotensin-aldosterone system (RAAS) as a significant biochemical hormonal axis and feedback mechanism in vasodilatory shock after they published the results of the Angiotensin II in High Output Shock Trial. Gleeson et al (8) showed in 2018 that renin appeared to be a much stronger and significant predictor of ICU mortality compared with lactate in a heterogenous shock population Jeyaraju et al (9) reported that renin kinetics are superior to lactate kinetics for predicting in-hospital mortality in critically ill patients with hypotension, with most being vasodilatory shock (most common diagnosis sepsis, also vasoplegia, acute respiratory distress syndrome [ARDS], liver failure) and those who had hypotension more than 6 hours while of vasopressors included. The bottom line in the previous investigations is that renin was a better marker of poor outcomes in comparison with concurrently measured lactate levels in critically ill ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* anticipated stay >24 hours
* signed informed consent by patient or next-of-kin.
* Septic shock patients, septic shock was defined as persistent hypotension (defined as the need for vasopressors to maintain mean arterial pressure ≥ 65 mm Hg, and a serum lactate level > 18 mg/dL [2 mmol/L] despite adequate volume resuscitation

Exclusion Criteria:

* chronic kidney disease stage IV/V (baseline eGFR (estimated glomerular filtration rate) <30ml/min/1.73m2),
* do not resuscitate order.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Septic shock patients, septic shock was defined as persistent hypotension (defined as the need for vasopressors to maintain mean arterial pressure ≥ 65 mm Hg, and a serum lactate level > 18 mg/dL [2 mmol/L] despite adequate volume resuscitation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-06-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Plasma renin levels at enrollment and after 24, 48, and 72 hours in septic shock patients | At enrollment and after 24, 48, and 72 hours.

SECONDARY OUTCOMES:
28 days mortality | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Khaled A. AbdelRahman, Assistant professor, Study Chair — Assiut University; Nagwa M. Ibrahim, Professor, Study Chair — Assiut University; Abualauon M. Abedalmohsen, Lecturer, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided